CLINICAL TRIAL: NCT05919238
Title: A Multicenter Open-label Phase 1 Trial to Evaluate Safety and Preliminary Efficacy of Endovascularly Applied Vascular Targeted Photodynamic Therapy (VTP) for Patients With Locally Advanced Unresectable Pancreatic Ductal Adenocarcinoma
Brief Title: Padeliporfin VTP Treatment for Unresectable Pancreatic Adenocarcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Impact Biotech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLIN2301 PNCM101
Record Dates: First submitted 2023-05-19; First posted 2023-06-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Locally Advanced Unresectable Pancreatic Adenocarcinoma
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Part B recruitment will be opened upon completion of Part A light dose escalation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Part A (Experimental): will be a monotherapy light dose escalation with single dose of Padeliporfin at light laser doses of 200, 400 and 600 mW/cm for 10 minutes.
  Part A will proceed with light dose escalation and will continue until the maximum tolerated light dose (MTD) and/or recommended phase 2 dose (RP2D) is defined.
  Interventions: Combination Product: Padeliporfin Vascular Targeted Photodynamic (VTP) therapy
- Part B (Experimental): will be a dose expansion part at MTD/RP2D dose level identified in Part A to further assess the safety, tolerability, and treatment effect of the MTD and/ or RP2D
  Interventions: Combination Product: Padeliporfin Vascular Targeted Photodynamic (VTP) therapy

INTERVENTIONS:
Combination Product: Padeliporfin Vascular Targeted Photodynamic (VTP) therapy — The laser light fiber with inflatable balloon to dam SMA blood flow during light illumination will be placed by an Interventional Radiologist in the SMA via a transfemoral artery approach. The balloon will be inflated to impede blood flow for total of 10 minutes during light illumination
  Other Names: Padeliporfin VTP

SUMMARY:
This is a prospective, multicenter, non-randomized, open label light dose escalation phase I trial to evaluate the safety and preliminary efficacy of Padeliporfin vascular targeted photodynamic therapy (VTP) applied via endovascular fiber placement within a dilatation catheter, through the target artery(superior mesenteric artery (SMA), celiac artery (CA) or common hepatic artery (CHA)). The investigators will evaluate safety and preliminary efficacy of Padeliporfin VTP administered endovascularly using light dose escalation.

DETAILED DESCRIPTION:
This is a prospective, multicenter, non-randomized, open label light dose escalation phase I trial to evaluate the safety and preliminary efficacy of Padeliporfin vascular targeted photodynamic therapy (VTP) applied via endovascular fiber placement within a dilatation catheter, through the the target artery(superior mesenteric artery (SMA), celiac artery (CA) or common hepatic artery (CHA)).The investigators will evaluate safety and preliminary efficacy of Padeliporfin VTP administered endovascularly using light dose escalation.

Study Intervention: Patients enrolled in the study will undergo endovascular VTP, using Padeliporfin (WST-11) activated via endovascular fiber placement through the target artery(superior mesenteric artery (SMA), celiac artery (CA) or common hepatic artery (CHA))., with intravenous administration of Padeliporfin at a fixed dose of 4 mg/kg of padeliporfin di-potassium, followed by total of 10 min illumination at 753 nm.

For light dose escalation (Part A), a 3+3 dose-escalation schema will be used. In a subsequent expansion phase (Part B), the optimal light dose as per light dose escalation, will be used in an additional cohort of patients to further evaluate preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

1Patient is 18 years of age and older 2. Patient is capable of giving written informed consent 3. Patients with a diagnosis of Stage III pancreatic ductal adenocarcinoma, cytologically or histologically confirmed per American Joint Committee on Cancer (AJCC) staging criteria 4. Patients have an unresectable tumor, evaluated as Stage III according to National Comprehensive Cancer Network (NCCN) guidelines resectability criteria, based on radiographic imaging or exploratory surgery as a locally advanced (LA) pancreatic ductal adenocarcinoma (PDAC) 5. Patients with LA PDAC located in the head/uncinate process of the pancreas 6. Patient with target artery solid tumor contact ˃180° for a total contact length up to 3cm, and with entire target artery internal diameter 5-10 mm. 7. All patients will be approved by a multi-disciplinary team (including medical oncologist, surgeon, interventional radiologist) as appropriate for endovascular VTP treatment. 8. Measurable disease as defined by the Response Evaluation Criteria in Solid Tumors according to RECIST 1.1 9. ECOG performance status ≤ 1 10. Life expectancy at least 6 months 11. No evidence of metastatic disease by CT scan chest, abdomen and pelvis performed within 28 days prior to treatment 12. Adequate organ system function including:

a. Absolute neutrophil count (ANC) ≥1500/mm3 without the use of hemopoietic growth factors within the 7 days before VTP treatment b. Absolute white blood cell count ≥3.0*109/L c. Hemoglobin at least 10g/dL d. Platelet count ≥75,000/mm3 e. International normalized ratio (INR) <1.5 unless the patient is receiving anticoagulation therapy, in which case a therapeutic INR is acceptable. Anticoagulation therapy with low- molecular-weight heparin whether medically indicated, is permitted. f. Creatinine clearance ≥60 mL/min using Cockcroft-Gault equation g. Amylase and lipase <1.5xULN h. ALT/AST ≤2.5*ULN and total bilirubin ≤2*ULN (benign hereditary hyperbilirubinemias, e.g., Gilbert's syndrome, are permitted, those patients must have total bilirubin <3 mg/dL).

13. Patient may have received prior neoadjuvant systemic therapy (chemotherapy and/or immunotherapy) 14. Patient with no prior external beam radiation therapy to the pancreas 15. Patient with prior attempted surgical resection is permitted 16. No comorbidities which would preclude access to the target artery by endovascular catheterization 17. Male or nonpregnant and nonlactating female aged ≥18 years

* Women of child-bearing potential (i.e., fertile, following menarche, and until becoming postmenopausal unless permanently sterile; permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) must test negative for pregnancy at the time of screening on the basis of a urine or serum pregnancy test.
* Postmenopausal women are defined as those who have had an absence of menstruation for at least 2 years.
* Female subjects of reproductive potential must agree to use two effective methods of birth control during the study and for 1 month after the last dose of study medication.
* Male subjects must agree to use condoms during the study and for 90 days after the last dose within the 7 days before VTP treatment of study medication.

Participant exclusion criteria

1. Metastatic (stage IV) disease
2. SMA originated not from aorta
3. Any anatomical variant or vascular abnormality that precludes safe placement of the balloon and device assembly in the target artery in the discretion of the principle investigator.
4. Hemodynamically significant moderate to severe atherosclerotic flow limiting changes of target vessel wall
5. Hemodynamically significant stenosis of the CA
6. Previous radiotherapy treatment for pancreatic cancer
7. Cystic component >= 25% the total volume of the tumor
8. Moderate to severe clinical ascites not controlled by medication detected by CT, ultrasound (US) or MRI;
9. Known additional malignancy that is progressing and/or requires active treatment.
10. Cardiac function: history of congestive heart failure or recent (within 6 months) myocardial infarction or ischemic event
11. Unable to receive or previously intolerant of moderate and/or deep sedation
12. Any other medical or social condition deemed by the investigator to be likely to interfere with a subject's ability to sign informed consent, cooperate, and participate in the study or that is likely to interfere with the interpretation of the results
13. Unwilling or unable to comply with study procedures and/or study visits
14. Receipt of prior definitive resection for pancreatic cancer
15. Pregnant and/or nursing
16. Active infection
17. Known hypersensitivity to iodine contrast
18. Receipt of concurrent investigational therapy or within 30 days of protocol initiation
19. Any other medical or psychiatric comorbidities, including decompensated heart failure, unstable angina or coronary artery disease or severe pulmonary disease, that, in the opinion of the study investigator, would make the patient a poor candidate for the study. Systemic chemotherapy treatment within at least 14 days prior to planned VTP. Preferred wash out period is 30 days.

21. VEGF-targeted therapy within 2 months prior to planned VTP treatment 22. Prohibited medication that could not be adjusted or discontinued prior to study treatment (See Section 16 for instructions) 23. Patients with photosensitive skin diseases or porphyria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety of endovascularly applied Padeliporfin VTP ablation | Day 30
  Safety of endovascularly applied Padeliporfin VTP ablation will be assessed using the CTCAE version 5.0. All adverse events (AEs) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) for being included in analyses.
Determination of the Maximum Tolerated Light Dose (MTD) and/or Recommended Phase 2 light dose (RP2D) in Part A | Day 30
  MTD is defined as the dose level associated with <33% of DLT-evaluable patients experiencing a DLT. If the MTD is reached, the RP2D will be defined as MTD. If the MTD is not reached, the RP2D will be selected based on integrated evaluation of safety and clinical benefit for all dose levels tested.

SECONDARY OUTCOMES:
Descriptive features of treatment response to ablation in tumor tissue based on pre- and post -VTP CT scans | Day 2
  Rate of resectability and downstaging (as per NCCN Clinical Practice Guidelines V1, May 4, 2023)
Tumor Response by CT scans | Day 30
  Based on CT scan according to RECIST 1.1
Tumor Response by CT scans | Day 60
  Based on CT scan according to RECIST 1.1

OTHER OUTCOMES:
Exploratory endpoints | 60 days
  Rate of resectability and downstaging will be evaluated by determining the percentage of patients who were initially deemed to have unresectable LA PDAC and following Padeliporfin VTP treatment, were subsequently deemed to have borderline resectable or resectable disease

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Abi-Jaoudeh, MD, Principal Investigator — University of California, Irvine
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - University of California Irvine, Irvine, California

IPD SHARING:
Plan to Share IPD: No